CLINICAL TRIAL: NCT02988362
Title: An Open-label, Randomized, Cross-over Study to Evaluate Pharmacokinetics and the Safety of HL068 16/10mg Compared to Candesartan 16mg and Amlodipine 10mg Co-administered in Healthy Male Volunteers.
Brief Title: Bioequivalence Study (Candesartan 16 mg and Amlodipine 10 mg)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HL068
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — candesartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Candesartan 16mg and Amlodipine 10mg (Experimental): Candesartan 16mg and Amlodipine 10mg
  Interventions: Drug: Candesartan 16mg and Amlodipine 10mg
- HL068 (Experimental): HL068(combination of Candesartan 16 mg and Amlodipine 10 mg)
  Interventions: Drug: HL068 16/10mg

INTERVENTIONS:
Drug: HL068 16/10mg — Candesartan 16mg and Amlodipine 10mg
  Arms: HL068
Drug: Candesartan 16mg and Amlodipine 10mg
  Arms: Candesartan 16mg and Amlodipine 10mg

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetics of HL068 (Candesartan 16 mg and Amlodipine 10mg) with coadministration of the two separate drugs in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer in the age between 19 and 55 years old.
* Body mass index (BMI) in the range of 18.5 to 27.0 kg/m2
* Understand the requirements of the study and voluntarily consent to participate in the study.

Exclusion Criteria:

* Previous history or present of clinically significant digestive , cardiovascular, respiratory, psychiatric, endocrine, hepatobiliary, renal disease.
* History of gastrointestinal disease or gastrointestinal surgery to affect drug absorption.
* Subjects with a hereditary problems, for example, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
* Subjects whose clinical laboratory test values are outside the accepted normal range. Especially, ASTor ALT >1.5 times of the Upper Normal Limit or total bilirubin > 1.5 times of the Upper Normal Limit
* Positive test results for Hepatitis B antibodies, Hepatitis C virus antibody, and Syphilis regain test
* Participation in any clinical investigation within 3 months prior to study drug administration
* Subjects with whole blood donation within 60 days or component blood donation within 30days or blood transfusion within 30days prior to the first dosing.
* SBP ≥ 140 mmHg or< 115 mmHg, DBP ≥ 90 mmHg or < 70 mmHg
* Caffeine > 400mg/day
* Alcohol > 30g/day
* Cigarette > 10 cigarettes/day.
* Subjects who are judged unsuitable by investigators

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2017-02-04 (Actual); Study Completion 2017-02-04 (Actual)

PRIMARY OUTCOMES:
AUCt | up to 72 hours
Cmax | up to 72 hours

SECONDARY OUTCOMES:
AUCinf | up to 72 hours
Tmax | up to 72 hours
t 1/2β | up to 72 hours
CL/F | up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Young-Ran Yoon, M.D, Ph.D, Principal Investigator — KYUNGPOOK NATIONAL UNIVERSITY HOSPITAL CLINICAL TRIAL CENTER

REFERENCES:
- [Derived] Lee HW, Kang WY, Jung W, Gwon MR, Yang DH, Kim EH, Cho K, Yoon YR, Seong SJ. Pharmacokinetics and bioequivalence of fixed-dose combination of candesartan cilexetil/amlodipine besylate (16/10 mg) versus coadministration of individual formulations in healthy subjects. Transl Clin Pharmacol. 2020 Jun;28(2):92-101. doi: 10.12793/tcp.2020.28.e8. Epub 2020 Jun 24. PMID 32656160